CLINICAL TRIAL: NCT00899093
Title: A Prospective, Longitudinal Study of YKL-40 in Patients With FIGO Stage III or IV Invasive Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Cancer Undergoing Primary Chemotherapy
Brief Title: YKL-40 in Serum Samples From Patients With Newly Diagnosed Stage III-IV Ovarian Epithelial, Primary Peritoneal Cavity, or Fallopian Tube Cancer Receiving Chemotherapy
Status: Terminated | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-0235; NCI-2009-01083 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000540250; GOG-0235 (Other: NRG Oncology); GOG-0235 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Fallopian Tube Adenocarcinoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Malignant Ovarian Brenner Tumor; Malignant Ovarian Clear Cell Tumor; Malignant Ovarian Endometrioid Tumor; Malignant Ovarian Mixed Epithelial Tumor; Malignant Ovarian Mucinous Tumor; Malignant Ovarian Neoplasm; Malignant Ovarian Serous Tumor; Malignant Ovarian Transitional Cell Tumor; Ovarian Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer; Undifferentiated Fallopian Tube Carcinoma; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Brenner Tumor; Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ancillary-Correlative (serum collection for YKL-40 and CA125): Patients undergo collection of serum samples for analysis of YKL-40 via ELISA and CA125 via chemiluminometric sandwich immunoassay at the following time-points: at baseline; prior to beginning each course of chemotherapy (courses 1-6); at completion of chemotherapy; every 3 months during years 1-2 post-chemotherapy; every 6 months during years 3-5 post-chemotherapy; every year during years 6-10 post-chemotherapy; and at time of disease recurrence or progression.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies chitinase 3-like 1 (cartilage glycoprotein-39) (YKL-40) in serum samples from patients with newly diagnosed stage III-IV ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer receiving chemotherapy. Studying samples of serum in the laboratory from patients receiving chemotherapy may help doctors learn more about the effects of chemotherapy on cells. It may also help doctors understand how well patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the ability of the YKL-40 serum marker to detect response or lack of response to primary chemotherapy in International Federation of Gynecology and Obstetrics (FIGO) stage III or IV invasive epithelial ovarian, primary peritoneal, or fallopian tube cancer.

II. To compare the predictive accuracy of YKL-40 with cancer antigen 125 (CA125).

SECONDARY OBJECTIVES:

I. To test the ability of the YKL-40 serum marker to detect recurrence of ovarian, primary peritoneal, or fallopian tube cancer in patients who are in first remission following primary chemotherapy.

II. To test the ability of the YKL-40 serum marker to predict poor risk patients with FIGO stage III or IV invasive epithelial ovarian, primary peritoneal, or fallopian tube cancer.

TERTIARY OBJECTIVES:

I. To explore alternative cut-off values for YKL-40 elevation in this large patient population.

II. To describe the variability of YKL-40 and CA125 measurements in patients receiving primary chemotherapy and in primary remission in a large patient population.

III. To describe the accuracy of YKL-40 coupled with CA125 measurements in predicting chemotherapy response, progression-free survival and overall survival.

OUTLINE:

Patients undergo collection of serum samples for analysis of YKL-40 via enzyme-linked immunosorbent assay (ELISA) and CA125 via chemiluminometric sandwich immunoassay at the following time-points: at baseline; prior to beginning each course of chemotherapy (courses 1-6); at completion of chemotherapy; every 3 months during years 1-2 post-chemotherapy; every 6 months during years 3-5 post-chemotherapy; every year during years 6-10 post-chemotherapy; and at time of disease recurrence or progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of FIGO stage III or IV invasive epithelial ovarian, primary peritoneal, or fallopian tube carcinoma who will receive primary chemotherapy for newly diagnosed disease; eligible histologic cell types include serous, mucinous, endometrioid, clear cell, transitional, mixed epithelial, undifferentiated, adenocarcinoma, not otherwise specified (NOS) and malignant Brenner tumor
* Patients who have undergone full surgical staging as described in the Gynecologic Oncology Group (GOG) Surgical Procedures Manual
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* The following histologic cell types are not eligible: carcinosarcoma (malignant mixed Mullerian tumor) and borderline epithelial tumors (low malignant potential, atypical proliferative)
* Patients with a current diagnosis of borderline epithelial ovarian tumor (formerly "tumors of low malignant potential") or recurrent invasive epithelial ovarian cancer treated with surgery only (such as those with stage IA or IB low grade lesions) are not eligible; patients with a prior diagnosis of a borderline tumor that was surgically resected and who subsequently develop an unrelated, new invasive epithelial ovarian or peritoneal primary cancer are eligible, provided that they have not received prior chemotherapy for any ovarian tumor
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded, unless all of the following conditions are met: stage not greater than IB; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other FIGO grade 3 lesions
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last five years or whose previous cancer treatment contraindicates this protocol therapy are excluded
* Patients who receive neoadjuvant chemotherapy prior to surgical staging
* Individuals with a diagnosis of rheumatoid arthritis, severe uncontrolled osteoarthritis, hepatic fibrosis or other active chronic inflammatory condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Newly Diagnosed Stage III-IV Ovarian Epithelial, Primary Peritoneal Cavity, or Fallopian Tube Cancer Receiving Chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2007-09; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
CA125 measurements | Up to 10 years
  The accuracy of each marker alone will be compared using area under the ROC curve, and assess which adds more predictive information when both are included in logistic regression.
Objective response using Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Up to 10 years
  In order to make a valid comparison between CA125 and YKL-40, in this study computed tomography (CT) criteria will be treated as the "gold standard" and whether changes in YKL-40 levels correlate with CT evidence as well as or better than changes in CA125 levels will be evaluated.
Time to disease progression using RECIST criteria | Up to 10 years
  Parallel statistical analyses of time to disease progression will also be conducted for patients who do not respond.
Time to tumor recurrence (relapse) | From study entry until disease recurrence, death or date of last contact, assessed up to 10 years
  Parallel analyses of the markers as predictors of time-to-relapse will be performed using survival-type regression methods such as the Cox proportional hazards model or a parametric maximum likelihood model. The total number of patients available for analysis of time to relapse is the number of patients who respond to treatment.
YKL-40 measurements | Up to 10 years
  YKL-40 will be compared to CA125 in terms of its ability to detect response to chemotherapy (during chemotherapy) and recurrence of disease (in remission). Serum YKL-40 behavior will also be assessed as a reflection of tumor histology, tumor grade, and tumor stage-all in comparison to CA125. The accuracy of each marker alone will be compared using area under the receiver operating characteristic (ROC) curve, and assess which adds more predictive information when both are included in logistic regression.

OTHER OUTCOMES:
Chemotherapy response | Up to 10 years
  As an exploratory analysis, the accuracy of YKL-40 coupled with CA125 measurements in predicting chemotherapy response will be described.
Optimal cut-off values for YKL-40 | Up to 10 years
  Optimal cut-off values for YKL-40 that subsequently can be used in clinical practice will be determined. Any statistical significance calculated for an optimized cut-off will adjust for the selection process, and any comparison with CA-125 will treat both markers in the same way.
Overall survival | From entry into the study to death or the date of last contact, assessed up to 10 years
  As an exploratory analysis, the accuracy of YKL-40 coupled with CA125 measurements in predicting overall survival will be described.
Progression-free survival | From study entry until disease progression, death or date of last contact, assessed up to 10 years
  As an exploratory analysis, the accuracy of YKL-40 coupled with CA125 measurements in predicting progression-free survival will be described.
Variability of CA125 measurements | Up to 10 years
  Linear statistical methods, such as a random effects model, will be used to assess the variability and correlation of CA125 over time in this population.
Variability of YKL-40 measurements | Up to 10 years
  Linear statistical methods, such as a random effects model, will be used to assess the variability and correlation of YKL-40 over time in this population.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bell-McGuinn, Principal Investigator — NRG Oncology
Locations (131):
- United States (131):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Highlands Oncology Group PA - Fayetteville, Fayetteville, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Northside Hospital, Atlanta, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Providence Medical Center, Kansas City, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Union Hospital of Cecil County, Elkton, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Island Gynecologic Oncology, Brightwaters, New York
  - New York Hospital Medical Center of Queens, Fresh Meadows, New York
  - Winthrop University Hospital, Mineola, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Knoxville Gynecologic Cancer Specialists PC, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin